CLINICAL TRIAL: NCT04808843
Title: Phase IV Study to Assess the Safety and Effectiveness of Dienogest (Visanne®) Amongst Indian Women With Endometriosis, in Real-world Clinical Practice: the VISAGE Study
Brief Title: A Study to Learn More About How Safe Dienogest is and How Well it Works Under Real World Conditions in Indian Women With Endometriosis
Acronym: VISAGE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19837
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis Associated Pelvic Pain
MeSH Terms: interventions — dienogest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dienogest: Patients with endometriosis who have been prescribed with Dienogest.
  Interventions: Drug: Dienogest (BAY86-5258, Visanne)

INTERVENTIONS:
Drug: Dienogest (BAY86-5258, Visanne) — Following the physicians' decision.

SUMMARY:
Endometriosis is a condition that affects women, usually during their reproductive years. In women with endometriosis, the tissue that normally covers the inside of the womb grows outside the womb. This can cause pain during their periods or during sex, and constant pain in the pelvis. Endometriosis can decrease a woman's quality of life. It also requires long-term treatment to control the symptoms.

The study drug, dienogest, has already been approved as a treatment for endometriosis associated pelvic pain. Sometimes, researchers continue studying a treatment after it has been approved to learn more about its safety.

In this study, the researchers want to learn more about any medical problems the patients have while taking dienogest. To answer this question, the researchers will collect the medical problems the patients have after taking dienogest and that may or may not be related to dienogest. These medical problems are also known as adverse events.

They will also collect information about the endometriosis associated pelvic pain. The pain measured with a standard rating scale called EAPP (endometriosis-associated pelvic pain) before treatment start and after 6 months of treatment will be compared.

The trial will include women with endometriosis associated pelvic pain whose doctors have decided to start treating them with dienogest. It will include about 160 women in India who are at least 18 years old.

All of the patients will take dienogest based on their doctor's instructions. They will then visit their study site 3 times over 6 months. At these visits, their doctors will ask them questions about how they are feeling and what medications they are taking. The doctors will do tests to measure the pain caused by the patients' endometriosis and any other symptoms. The doctors will also do physical examinations and check the patients' overall health.

ELIGIBILITY:
Inclusion Criteria:

* Female patients in India at least 18 years of age
* Clinical or surgical diagnosis of endometriosis: Clinical diagnosis by suggestive symptoms and positive finding in imaging study (Chocolate cyst)
* Patients diagnosed with endometriosis associated pelvic pain who have not been previously treated with Dienogest
* Decision to initiate treatment with Dienogest was made as per investigator's routine treatment practice
* Signed informed consent

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice
* Contra-indications according to the local summary of product characteristics (SPC)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indian female patients diagnosed with endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events that occur during treatment with Dienogest | 6 months
  Will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system

SECONDARY OUTCOMES:
Change in endometriosis associated pelvic pain | 6 months
  Measured by Numerical Rating Scale (NRS) on an 0-10 EAPP (Endometriosis Associated Pelvic Pain) NRS with "absence of pain" corresponding to the value "0" and "unbearable pain" corresponding to the value "10".

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, India

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.